CLINICAL TRIAL: NCT01993433
Title: A Randomized, Double-blind, Vehicle Controlled Study of the Safety and Efficacy of Topical DRM02 in Subjects With Plaque Psoriasis
Brief Title: A Safety and Efficacy Study of DRM02 in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRM02-PSO02
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRM02 (Experimental): DRM02 Topical Gel, 0.25%
  Interventions: Drug: DRM02
- Vehicle (Placebo Comparator): DRM02 Topical Gel, Vehicle
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: DRM02
  Arms: DRM02
Other: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine whether DRM02 is safe and effective in the treatment of plaque psoriasis when applied twice daily for 6 weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, within-subject control, study enrolling 20 subjects with plaque psoriasis and designed to assess the safety, tolerability, and preliminary efficacy of DRM02.

Safety will be assessed during the study, through adverse events, local skin responses, urinalysis, serum chemistry and hematology laboratory testing, physical examination and vital signs.

Preliminary efficacy will be assessed through the Physician's Lesion Assessment (PLA) and the Severity of Psoriasis Area Severity Index (PASI) from only the two plaques identified at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 70 years of age.
* Plaque-type psoriasis with two lesions of similar size and have an identical score of at least 6 but no more than 8 on the sum of the individual components of the Severity of Psoriasis Area Severity Index (PASI) at the Target Lesion scale.
* Male or non-pregnant, non-lactating females.
* Signed informed consent.

Exclusion Criteria:

* Subjects who have extensive, and/or 'inverse', and/or exfoliative psoriasis.
* Subjects who have taken any systemic treatment for psoriasis within the 4 weeks prior to baseline.
* Prior or concomitant use of topical treatments for psoriasis to within 10 cm of the target lesion within the 4 weeks prior to baseline.
* Use of Enbrel within the 4 weeks prior to baseline.
* Psoralen & ultraviolet A therapy (PUVA) or the use of ultraviolet B (UVB) therapy and/or excessive or prolonged exposure to ultraviolet light within the 4 weeks prior to baseline.
* Use of Humira or Remicade within the 3 months prior to baseline.
* Use of Stelara within the 6 months prior to baseline.
* Subjects who have taken oral retinoids for psoriasis within the 6 months prior to baseline.
* Subjects who have poor skin condition within 5 cm of the target lesion.
* Subjects who are current drug or alcohol abusers; have a history of immunodeficiency disease or are a poor medical risk because of other systemic diseases or active uncontrolled infections.
* Subjects with an unstable medical condition or a medical condition not adequately controlled with standard medical therapy.
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 30 days
* Subjects who have a clinically significant laboratory value at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Physician's Lesion Assessment | Week 6

SECONDARY OUTCOMES:
Physician's Lesion Assessment | From baseline to weeks 0, 1, 2, 3, 4 and 6
PLA dichotomized into "success" and "failure" | Week 6

OTHER OUTCOMES:
Severity of Target Lesion PASI scores | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Beth Zib, Study Director — Dermira, Inc.
Locations (2):
- Canada (2):
  - Clinique Médicale Dr Isabelle Delorme, Drummondville, Quebec
  - Innovaderm Research, Inc, Montreal, Quebec